CLINICAL TRIAL: NCT03863002
Title: Mesenchymal Stem Cell Transplantation for Acute-on-Chronic Liver Failure
Brief Title: Safety and Efficacy of Mesenchymal Stem Cell Transplantation for Acute-on-Chronic Liver Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Weikai Bioeng., Ltd. (Industry)
Collaborators: Tianjin Nankai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tianjin Weikai Bioeng., Ltd
Record Dates: First submitted 2019-02-18; First posted 2019-03-05 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2018-04

CONDITIONS: Liver Failure, Acute on Chronic
Keywords: mesenchymal stem cell
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Masking Description: both participants and the study team are unblinded to the treatment allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Treatment (No Intervention): Standard Medical Treatment (SMT): All patients received SMT, including nutritional supplementation; administration of human serum albumin (serum albumin <30 g/L), fresh frozen plasma (200-400 mL/day until the INR was <1.5), S-adenosylmethionine (1.0 g/day); or anti-virus treatment for hepatic viruses-related cases, and appropriate treatment for complications such as infections (including of the respiratory tract, urinary tract, biliary tract, and digestive tract and spontaneous peritonitis), encephalopathy, gastrointestinal bleeding, and hepatorenal syndrome [HRS]).
- Mesenchymal Stem Cell (Experimental): Mesenchymal Stem Cell (MSC): The MSC group received infusions of 1.0 to 10x10^5cells/kg MSCs through the peripheral vein once a week for 4 weeks, in addition to SMT.
  Interventions: Biological: Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Mesenchymal Stem Cell — Mesenchymal stem cell transplantation via peripheral vein: 1.0-10x10^5 MSCs/kg body weight administered via peripheral vein at week 0, 1, 2, 3 weeks
  Arms: Mesenchymal Stem Cell

SUMMARY:
Safety and Efficacy of Mesenchymal Stem Cell Transplantation for Acute-on-Chronic Liver Failure

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (ACLF) which occurs in patients with chronic liver disease, is a serious live-threatening disease. Currently, the clinical management, such as liver protection, anti-virus medicine, and artificial liver support, has not significantly improve the outcomes, the mortality still remains over 50%. Liver transplantation is the only effective treatment of ACLF, but this therapy is limited by the shortage of donor organs, potential surgical complications, immunological rejection and high medical costs. Mesenchymal stem cell (MSC) is one of adult stem cells, which has been suggested to play a role in amelioration of liver disease, such as: trans-differentiation of MSCs into hepatocytes, immunomodulation, inhibition of fibrosis development, protective effects on hepatic cell and restoration of hepatic cell proliferation capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Meeting the definition of ACLF: patients with previously diagnosed or undiagnosed chronic liver disease acute decompensated within 4 weeks; significant GI symptom as such fatigue, jaundice; serum total bilirubin [TBil] ≥10 X the upper limit of normal; coagulopathy (international normalized ratio [INR] ≥1.5 or prothrombin activity [PTA] <40%); complicated within 4 weeks by ascites and/or encephalopathy as determined by physical examination.
3. Model for End-Stage Liver Disease (MELD) scores ranging 17-30, (MELD(i) = 0.957 × ln(Cr) + 0.378 × ln(bilirubin) + 1.120 × ln(INR) + 0.643);
4. Chronic liver disease with definitive etiology such as viral hepatitis, alcohol liver disease, drug induced liver injury or autoimmune liver diseases
5. Body weight ≥50kg

Exclusion Criteria:

1. Serious complications in the previous 2 months (e.g., gastrointestinal bleeding: hemoglobin below 90g/L, serious infection such as sepsis, ascites ultrafiltration, and/or dialysis);
2. Malignant jaundice induced by obstructive jaundice or hemolytic jaundice;
3. Hepatocellular carcinoma (HCC) diagnosed by radiologic imaging and/or alpha fetoprotein (AFP);
4. Tumor diagnosed by ultrasound, CT, MR examination;
5. Moderate or severe chronic heart failure (NYHA III-IV), renal replacement therapy, severe chronic pulmonary disease (GOLD III-IV)
6. Extrahepatic cholestasis
7. Hepatic, portal and splenic vein thrombosis diagnosed by doppler ultrasound
8. Artificial liver support
9. Previous liver transplantation
10. Drug abuse in the past 5 years;
11. Mental disorders and/or has a family history of mental disorder.
12. HIV infection
13. Pregnant or breast-feeding females
14. Highly allergic
15. Patients can not cooperate or mobility
16. Enrolled in other clinical trials with 3 months
17. Patients who can not provide prior informed consent or refusal to participate

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
survival rate | 72 weeks after treatment
  Number of participants alive

SECONDARY OUTCOMES:
Adverse reactions | Week 1, 2, 4, 8, 12, 24, 36, 48
  Number of participants with adverse reactions (e.g. fever, rash, and diarrhea )
White blood cell | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of white blood cell count
Platelet | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of platelet count
Hemoglobin | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of hemoglobin level
Creatinine | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of creatinine level as a surrogate marker of liver function
ALT | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of alanine aminotransferase (ALT) level as a marker of liver function
ALB | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of albumin (ALB) level as a maker of liver function
TBil | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of total Bilirubin (TBil) level as a marker of liver function
INRs | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of international normalized ratio (INRs) level as a marker of liver function
AFP | Week 1, 2, 4, 8, 12, 24, 36, 48
  Change of alpha fetoprotein (AFP) level as a marker of liver function
MELD scores | Week 1, 2, 4, 8, 12, 24, 36, 48
  Model for End-Stage Liver Disease (MELD) score for assessing the severity of chronic liver disease is measured as absolute change to baseline score
Tumor formation | Week 1, 2, 4, 8, 12, 24, 36, 48
  Number of participants with hepatocellular carcinoma or extrahepatic malignant tumors
Liver failure-associated serious complications | Week 1, 2, 4, 8, 12, 24, 36, 48
  Number of participants with liver failure-associated serious complications, such as infections, encephalopathy, gastrointestinal bleeding and HRS

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Weikai Bioeng., Ltd., Tianjin, Tianjin Municipality, China